CLINICAL TRIAL: NCT03688087
Title: Study of Program Interest "Bouge" to Improve the Daily Physical Activity and Tolerance in Processings Treatment of Pregnant Women
Brief Title: Study of Programm Interest 'Bouge' to Improve the Daily Physical Activity at the Pregnant Women.
Acronym: BOUGE GROSSESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BOUGE GROSSESSE (29BRC17.0108)
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Physical Activity; Pregnant; Mobile Health Apps
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Smartphone application "placebo"
  Interventions: Device: Smartphone application "placebo"
- "Bouge" (Active Comparator): Smartphone equipped with the application "Bouge"
  Interventions: Device: Smartphone equipped with application "bouge" = Coach group

INTERVENTIONS:
Device: Smartphone application "placebo" — Strategy based on smartphone application "placebo"
  Arms: placebo
Device: Smartphone equipped with application "bouge" = Coach group — Strategy based on smartphone application "bouge"
  Arms: "Bouge"

SUMMARY:
Evaluate the "Bouge" digital program (smartphone application) to increase the daily physical activity of pregnant patients beguining at 15 SA

DETAILED DESCRIPTION:
Controlled, randomized, open, prospective, multicentric study, 250 pregnant patients aged between 18 and more, with 14 weeks of amenorrhea, possessing a smartphone, will be recruited and randomized into two groups:

125 in the control group (smartphone application "placebo" = number of steps) 125 will be equipped with the application "Bouge" = coached group

For three months, the patients do their daily physical activity. The "coached" group, through the smartphone application "Bouge", receives computer coaching to increase their physical activity (no direct medical intervention, only notifications and computer pusch).

The control group is not coached by the application (simple display of the number of step)

ELIGIBILITY:
Inclusion Criteria:

Pregnant <14 weeks of amenorrhea Must have a compatible smartphone

Exclusion Criteria:

Multiple pregnancies Pre-existing pregnancy-related diseases Pregnancy complicated History of peripheral arterial disease History of IUGR History of cone biopsy History of delivery hemorrhage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-10-22 (Estimated); Study Completion 2018-10-22 (Estimated)

PRIMARY OUTCOMES:
Increased daily physical activity (number of steps) using the smartphone application "BOUGE" | 12 Weeks
  The objective is an increase of 2000 steps daily between J 1 and J 90 (an increase of 10 000 steps between S1 and S 12)

SECONDARY OUTCOMES:
sleep, | 12 Weeks
  Scale Spiegel
Well being | 12 Weeks
  Scale OMS
- lumbago | 12 Weeks
  Scale EIFEL

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Clinique KERAUDREN, Brest
  - CHRU de Brest, Brest
  - CH de Morlaix, Morlaix
  - Chic Quimper, Quimper

REFERENCES:
- [Derived] Muller M, James P, Merviel P, Saraux A, Guillodo Y, Kerlan V, Bouee S, Nowak E, Morgant R, Communier-Courtois E. A smartphone coaching program ("Bouge Grossesse") improves daily physical activity in pregnant women. J Gynecol Obstet Hum Reprod. 2026 Feb;55(2):102847. doi: 10.1016/j.jogoh.2024.102847. Epub 2024 Sep 12. PMID 39277170